CLINICAL TRIAL: NCT04206982
Title: MARSHALL Bundles Elimination, Pulmonary Veins Isolation and Lines Completion for ANatomical Ablation of Persistent Atrial Fibrillation Versus Pulmonary Veins Isolation: The MARSHALL PLAN Monocentric Trial
Brief Title: MARSHALL PLAN Vs. Pulmonary Veins Isolation Monocentric Trial
Acronym: PLAN-MARSHALL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2019/08
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation
Keywords: Persistent atrial fibrillation; Pulmonary vein isolation; Catheter ablation; Ethanolisation; Ligament of Marshall
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: The Marshall Plan is a prospective randomized, parallel-group, monocentric clinical trial of superiority.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Marshall Plan arm (Experimental): Patients will undergo (1) the destruction of Marshall bundles by ethanol infusion followed by ablation of the distal coronary sinus bundles, the ridge and the saddle; (2) the standard pulmonary veins sleeves isolation; (3) and finally the ablation of the mitral, the roof, and the cavo-tricuspid isthmus.
  Interventions: Procedure: Destruction of Marshall bundles; Procedure: Pulmonary veins isolation; Procedure: Linear ablation in the left and right atria
- Pulmonary vein isolation arm (Active Comparator)
  Interventions: Procedure: Pulmonary veins isolation

INTERVENTIONS:
Procedure: Destruction of Marshall bundles — Destruction of Marshall bundles by ethanol 96% infusion (2 separate injections of 5ml on 1 minute each) followed by ablation of the distal coronary sinus bundles, the ridge and the saddle.
  Arms: Marshall Plan arm
Procedure: Pulmonary veins isolation — Achievement of a wide disconnection of the right and left pulmonary veins.
Procedure: Linear ablation in the left and right atria — Ablation of the mitral, the roof, and the cavo-tricuspid isthmus.
  Arms: Marshall Plan arm

SUMMARY:
In ablation strategy for persistent Atrial Fibrillation (PsAF), ablation limited to Pulmonary Vein (PV) isolation is the most straightforward approach but the result give only 50% of arrhythmia free follow-up. Substrate modification strategies have failed to demonstrate their superiority with variable reported success rate. The Marshall network is a highly arrhythmogenic structure that has not been incorporated in current ablation strategies. The investigators sought to investigate a new ablation strategy that target systematically the vein of Marshall by ethanol infusion. This step is integrated in a new ablation strategy consisting in a global anatomical substrate based ablation including PV isolation and left atrial linear ablation (Marshall-Plan).

The main objective of this study is to compare the 12 month freedom from any arrhythmia (Atrial Fibrillation (AF)/Atrial Tachycardia (AT)) between the Marshall-Plan approach and the PV isolation approach.

DETAILED DESCRIPTION:
Ablation strategy for persistent AF besides pulmonary vein isolation remains controversial. Indeed, two approaches have prevailed over the past two decades "cox-maze" strategy and mapping of the left atrium but both methods have failed to decrease AF recurrences (as shown by the clinical trial STAR AF 2). Two studies have demonstrated that the ligament of Marshall (LOM) could be the source of focal activities, the substrate of reentries and a strong parasympathetic modulator. For these reasons, LOM may represent a major target in AF treatment besides PV isolation. Nevertheless, conventional ablation techniques do not ensure the complete destruction of Marshall's musculature and parasympathetic ganglia that surround it, largely isolated by a sheath of adipose tissue. To overcome this technical limitation, LOM elimination can be achieved by alcohol injection into the vein of Marshall.The investigator innovative approach called Marshall Plan will then consists in 3 steps: 1) the destruction of Marshall bundles by ethanol infusion followed by the ablation of the distal Coronary Sinus (CS) bundles, the ridge and the saddle; 2) the standard PV isolation; 3) and finally ablation of the mitral line, the roof and of the cavo-tricuspid isthmus, main causes of recurrence in atrial flutter.

Before ablation procedure patients will be randomized in 2 arms: Marshall Plan (treatment arm) or pulmonary vein isolation (control arm). Patients will be followed at 3, 6, 9 and 12 months in-office visits or hospitalization. Patients will have different tests: electrocardiogram (ECG), cardiac echography, stress test, 24hours Holter and transtelephonic ECG monitor with weekly transmitted ECG and at any time in case of symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of both genders
* Suitable candidate for catheter non-emergent mapping and ablation of atrial fibrillation defined as:

  * History of symptomatic persistent atrial fibrillation in the past year documented by ECG AND
  * Treatment failure by at least one class of anti-arrhythmic medications (I-IV) (intolerance or recurrence of symptomatic AF)
* Patient affiliated or beneficiary of social security scheme
* Free, informed and written consent signed by the participant and the principal investigator (at least at the inclusion date and before all exams required for the clinical research)
* Effective contraception for women of childbearing potential

Exclusion Criteria:

* Minor
* Prior left atrial heart ablation procedure
* Documented left atrial thrombus or another abnormality which precludes catheter introduction
* Contraindication to anticoagulation therapy (heparin, warfarin, or Novel Oral Anticoagulant (NOAC)
* Contraindication to iodinated contrast product XENETIX® (iobitridol hypersensitivity or at one of these excipients, history of major immediate reaction or cutaneous reaction to XENETIX® infusion, thyrotoxicosis)
* Hypersensitivity to ethanol
* Unstable angina or ongoing myocardial ischemia
* Myocardial infarction within 3 months prior to inclusion
* Congenital heart disease, where the underlying abnormality increases the ablation risk
* Pulmonary hypertension (pulmonary arterial hypertension > 50 mmHg)
* Severe uncontrolled systemic hypertension with systolic blood pressure (SBP) > 200 mm Hg within 30 days prior to inclusion
* Severe bleeding, clotting or thrombotic disorder
* Left atrial diameter > 60 mm (parasternal view)
* Hypertrophic cardiomyopathy defined by a left ventricular septum thickness > 1.5 cm
* Pregnant, parturient or nursing women
* Unable or unwilling to provide written informed consent
* Patient detained by judicial or administrative order
* Patient under psychiatric care
* Patient admitted in a social or healthcare establishment for any purpose other than the research
* Subject to a legal protection order (guardianship, patient under legal protection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Recurrence of AF or AT greater than 30 seconds with or without antiarrhythmic medications. | 12 months
  Recurrence rate (percentage) of AF or AT > 30 seconds after the blanking period of 3-months post ablation, at 12 months with or without antiarrhythmic medications. Recurrences will be identified through transtelephonic ECG monitor with weekly transmitted ECG and at any time in case of symptoms.

SECONDARY OUTCOMES:
Recurrence of AF greater than 30 seconds | 12 months
  Recurrence rate (percentage) of AF greater than 30 seconds after the blanking period of 3-months post procedure at 12 months. It will be identified through transtelephonic ECG monitor with weekly transmitted ECG and at any time in case of symptoms.
Recurrence of AF or AT greater than 30 seconds without antiarrhythmic medications | 12 months
  Recurrence rate (percentage) of AF or AT > 30 seconds after the blanking period of 3-months post ablation, at 12 months without antiarrhythmic medications. Recurrences will be identified through transtelephonic ECG monitor with weekly transmitted ECG and at any time in case of symptoms.
Rate of patients under antiarrhythmic medications | 12 months
  Percentage of patients
Number of patients with repeat procedures | 12 months
  Number of patients
Rate of periprocedural complications | 12 months
  Percentage of transient ischemic attack or stroke, cardiac tamponade, atrio-oesophageal fistula, pericarditis, complications at access site (hematoma, arteriovenous fistula, pseudoaneurysm).
AF discontinuation rate during procedure | 12 months
  Percentage of AF discontinuation
Per-procedure AF / AT inducibility rate | 12 months
  Percentage of per-procedure AF / AT inducibility
Mitral line block rate | 12 months
  Percentage of mitral line block according to consensus block criteria
Radiofrequency duration necessary for pulmonary veins isolation | 12 months
  Duration measured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas DERVAL, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Bordeaux University Hospital, Pessac, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valderrabano M, Chen HR, Sidhu J, Rao L, Ling Y, Khoury DS. Retrograde ethanol infusion in the vein of Marshall: regional left atrial ablation, vagal denervation and feasibility in humans. Circ Arrhythm Electrophysiol. 2009 Feb;2(1):50-6. doi: 10.1161/CIRCEP.108.818427. PMID 19756206
- [Derived] Derval N, Tixier R, Duchateau J, Bouteiller X, Loock T, Denis A, Chauvel R, Bouyer B, Arnaud M, Yokoyama M, Kowalewski C, Monaco C, Ascione C, Sacher F, Hocini M, Jais P, Haissaguerre M, Pambrun T. Marshall-Plan Ablation Strategy Versus Pulmonary Vein Isolation in Persistent AF: A Randomized Controlled Trial. Circ Arrhythm Electrophysiol. 2025 May;18(5):e013427. doi: 10.1161/CIRCEP.124.013427. Epub 2025 May 20. PMID 40392905